CLINICAL TRIAL: NCT05592470
Title: The Copper Metabolism MURR1 Domain 7 (COMMD7) Gene Expression in Acute Lymphoblastic Leukemia
Brief Title: commd7 Gene Expression in ALL
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Marwa Saad Mohamed Mahrous, AssuitU, Assiut University
Other Study IDs: commd7 gene expression in ALL
Record Dates: First submitted 2022-10-20; First posted 2022-10-24 (Actual); Last update posted 2022-10-24 (Actual); Status verified 2022-09

CONDITIONS: ALL
Keywords: COMMD7 , ALL

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- PATEINTS: 51 patients newly diagnosed with acute lymphoblastic leukemia
  Interventions: Diagnostic Test: Reverse transcription-quantitative polymerase chain reaction (RT-qPCR).
- controls: 51 normal persons
  Interventions: Diagnostic Test: Reverse transcription-quantitative polymerase chain reaction (RT-qPCR).

INTERVENTIONS:
Diagnostic Test: Reverse transcription-quantitative polymerase chain reaction (RT-qPCR). — Reverse transcription-quantitative polymerase chain reaction on bone marrow aspirates to detect The expression pattern of COMMD7 gene in acute lymphoblastic leukemia

SUMMARY:
* study the expression pattern of COMMD7 gene in acute lymphoblastic leukemia.
* investigate correlation between the expression level of COMMD7 gene with other diagnostic parameters and prognosis in ALL .

DETAILED DESCRIPTION:
Acute lymphoblastic leukemia (ALL) is a neoplastic disorder of lymphoid progenitor cells characterized by diverse cytogenetic and molecular abnormalities with peaks of prevalence for 2-5-year-old patients and those older than 50. Treatment strategies using risk-adapted chemotherapy cure more than 80% of childhood cases, but around 20 to 30% relapse developing serious complications including death.( 1) In the past decade, the available treatments for patients with acute lymphoblastic leukemia (ALL) have rapidly expanded, in parallel with an increased understanding of the genomic features that impact the disease biology and clinical outcomes.(2) The copper metabolism MURR1 domain (COMMD) protein family involved in tumor development and progression in several types of human cancer, but little is known about the function of COMMD proteins in hematological malignancy. (3) COMMD7, a member of the COMMD, which is located on chromosome 20q11.21, has been reported associated with tumor progression in human solid cancers [4]. COMMD7 is overexpressed in pancreatic ductal adenocarcinoma (PDAC) cells, associated with poor prognosis. [5]. Another study revealed that COMMD7-overexpressed hepatocellular carcinoma (HCC) cells promoted the proliferation of naïve HCC cells (6) A recent study was found that high expression of COMMD7 is a potential biomarker for adverse outcomes and poor prognosis in AML. (7)

. However, to date, the expression of COMMD7 in acute lymphoblastic leukemia and its prognostic value remain unclear.

ELIGIBILITY:
Inclusion Criteria:

* Patients newly diagnosed with acute lymphoblastic leukemia , male or female at any age.

Exclusion Criteria:

* history of anti-neoplastic therapy, such as chemotherapy or radiotherapy.
* Any other types of cancers.
* Any clinically systemic acute or chronic inflammatory disease/s within one months.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The required sample size will be 102 subject (51 newly diagnosed patients with ALL and 51 controls )
Sampling Method: Probability Sample
Enrollment: 102 (Estimated)
Dates: Start 2022-11 (Estimated); Primary Completion 2024-04 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
The expression pattern of COMMD7 gene in acute lymphoblastic leukemia | BASELINE
  Reverse transcription-quantitative polymerase chain reaction (RT-qPCR) TO DETECT EXPRESSION pattern in ALL

SECONDARY OUTCOMES:
Correlation between the expression level of COMMD7 GENE with other diagnostic parameters and prognosis in ALL | baseline

REFERENCES:
- [Background] Garza-Veloz I, Martinez-Fierro ML, Jaime-Perez JC, Carrillo-Sanchez K, Ramos-Del Hoyo MG, Lugo-Trampe A, Rojas-Martinez A, Gutierrez-Aguirre CH, Gonzalez-Llano O, Salazar-Riojas R, Hidalgo-Miranda A, Gomez-Almaguer D, Ortiz-Lopez R. Identification of differentially expressed genes associated with prognosis of B acute lymphoblastic leukemia. Dis Markers. 2015;2015:828145. doi: 10.1155/2015/828145. Epub 2015 Feb 24. PMID 25802479
- [Background] Short NJ, Kantarjian H, Jabbour E. Optimizing the treatment of acute lymphoblastic leukemia in younger and older adults: new drugs and evolving paradigms. Leukemia. 2021 Nov;35(11):3044-3058. doi: 10.1038/s41375-021-01277-3. Epub 2021 Jun 25. PMID 34172894
- [Background] Bartuzi P, Hofker MH, van de Sluis B. Tuning NF-kappaB activity: a touch of COMMD proteins. Biochim Biophys Acta. 2013 Dec;1832(12):2315-21. doi: 10.1016/j.bbadis.2013.09.014. Epub 2013 Sep 29. PMID 24080195
- [Background] Burstein E, Hoberg JE, Wilkinson AS, Rumble JM, Csomos RA, Komarck CM, Maine GN, Wilkinson JC, Mayo MW, Duckett CS. COMMD proteins, a novel family of structural and functional homologs of MURR1. J Biol Chem. 2005 Jun 10;280(23):22222-32. doi: 10.1074/jbc.M501928200. Epub 2005 Mar 30. PMID 15799966
- [Background] You N, Li J, Gong Z, Huang X, Wang W, Wang L, Wu K, Zheng L. COMMD7 functions as molecular target in pancreatic ductal adenocarcinoma. Mol Carcinog. 2017 Feb;56(2):607-624. doi: 10.1002/mc.22520. Epub 2016 Jul 8. PMID 27350032
- [Background] You N, Li J, Huang X, Wu K, Tang Y, Wang L, Li H, Mi N, Zheng L. COMMD7 promotes hepatocellular carcinoma through regulating CXCL10. Biomed Pharmacother. 2017 Apr;88:653-657. doi: 10.1016/j.biopha.2017.01.046. Epub 2017 Jan 29. PMID 28142122
- [Background] Li K, Chen L, Zhang H, Wang L, Sha K, Du X, Li D, Zheng Z, Pei R, Lu Y, Tong H. High expression of COMMD7 is an adverse prognostic factor in acute myeloid leukemia. Aging (Albany NY). 2021 Apr 23;13(8):11988-12006. doi: 10.18632/aging.202901. Epub 2021 Apr 23. PMID 33891561